CLINICAL TRIAL: NCT07165990
Title: Produce Rx in High Risk Pregnant Mothers at Harris Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0734 (phase 3)
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Methods; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Food is Medicine (FIM) Intervention plus Standard of Care (Experimental)
  Interventions: Behavioral: Food is Medicine (FIM) Intervention; Behavioral: Standard of Care
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Food is Medicine (FIM) Intervention — Intensive intervention phase - this phase starts at enrollment (<=14 weeks) through 28 weeks of gestation (or at the time of GDM diagnostic test) and women i) receive a bi-weekly home delivery of a "mixed box" consisting of fresh produce, lean protein, and whole grains combined with culinary medicine-based nutrition education available in English and Spanish.
  Maintenance phase - this phase starts at 29 weeks through 12 weeks postpartum, and women will receive biweekly deliveries of about 10-15 pounds of fresh produce (8-10 different kinds of produce) plus standard nutrition education. The box will be curated for prenatal nutrients needs and following American Diabetes Association guidelines.
  Arms: Food is Medicine (FIM) Intervention plus Standard of Care
Behavioral: Standard of Care — Standard medical care provided at Harris Health for high-risk pregnant women, plus a voucher equal to the value of the produce and meals provided in the Food is Medicine (FIM) Intervention.

SUMMARY:
The purpose of this study is to assess the effectiveness of a "Food is Medicine" (FIM) intervention on incidence of gestational diabetes mellitus (GDM) among pregnant women at risk for GDM within the Harris Health system.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women receiving care at Harris Health clinics
* Medicaid eligible or receiving Medicaid
* <=14 weeks gestation at the time of the first prenatal visit and study enrollment
* meet the ACOG criteria for early screening for GDM (have a BMI of 30 or greater and at least one additional ACOG-designated risk factor for GDM from the following: Age > 35 years; Black, Hispanic, Native American, Asian American or Pacific Islander ethnicity; history of GDM in prior pregnancy; A1c level > 5.7 & < 6.4; history of hypertension, pregnancy hypertension, heart disease, HIV, high triglycerides, polycystic ovarian syndrome; Immediate family member (parent or sibling) has had diabetes)
* fall within the study delivery radius

Exclusion Criteria:

* report existing or pregestational T2DM
* have hemoglobin A1c>=7
* are prescribed insulin therapy or metformin upon first screening

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with gestational diabetes mellitus (GDM) | 24-28 weeks gestational age (about 10-12 weeks after start of the intervention)

SECONDARY OUTCOMES:
Number of participants with hypertensive disorders of pregnancy | 24-28 weeks gestational age (about 10 weeks after start of the intervention)
Number of infants with macrosomia at birth | at the time of birth
Number of infants with pre-term birth | at the time of birth
Number of infants born via C-section | at the time of birth
Change in Hemoglobin A1c levels | at the time of the first prenatal visit, at the time of birth

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No